CLINICAL TRIAL: NCT00492687
Title: A Phase II Pilot Trial of Radiation Therapy With Concurrent and Adjuvant Temozolomide, Tamoxifen and Carboplatin (T2C) in the Treatment of Patients With Primary Central Nervous System Malignant Gliomas
Brief Title: Radiation Therapy, Temozolomide, Tamoxifen, and Carboplatin in Treating Patients With Malignant Gliomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Diego Pacific Oncology & Hematology Associates (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000551555; POHA-0601
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma; adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Glioblastoma; Gliosarcoma | interventions — Carboplatin; Tamoxifen; Temozolomide; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: tamoxifen citrate
Drug: temozolomide
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Tamoxifen may make tumor cells more sensitive to radiation therapy and chemotherapy. Giving radiation therapy together with temozolomide, tamoxifen, and carboplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving radiation therapy together with temozolomide, tamoxifen, and carboplatin works in treating patients with malignant gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression-free and overall survival of patients with supratentorial malignant gliomas (WHO grade III or IV) receiving radiotherapy with concurrent and adjuvant temozolomide, tamoxifen citrate, and carboplatin.
* Determine the acute and delayed treatment-related toxicities in these patients.
* Determine tumor response in patients with postoperative measurable disease.

OUTLINE: This is an open-label, pilot study.

* Induction therapy: Patients receive oral temozolomide twice daily and oral tamoxifen citrate twice daily on days 1-42 and carboplatin IV over 60 minutes on days 1, 8, 15, 22, 29, and 36. Patients also receive radiotherapy on days 1-5 in weeks 1-6.
* Consolidation therapy: Beginning 4 weeks after the completion of induction therapy, patients receive temozolomide, tamoxifen citrate, and carboplatin as in induction therapy. Treatment repeats every 8 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme and/or anaplastic astrocytoma

  * Supratentorial tumor
  * No well-differentiated astrocytoma or glioma with oligodendroglial component
  * No multifocal glioma
* Has undergone surgery within the past 6 weeks
* No recurrent glioblastoma multiforme

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Neurological functional status 0-2
* Life expectancy > 12 weeks
* ANC ≥ 1,200/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Blood urea nitrogen ≤ 1.5 times ULN
* Total and direct bilirubin ≤ 3 times ULN
* AST and ALT ≤ 3 times ULN
* Alkaline phosphatase ≤ 3 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study completion
* No other malignancies within the past 3 years, except for carcinoma in situ of the cervix or nonmelanoma skin cancer
* No acquired immune deficiency syndrome (AIDS)
* No major medical illness or psychiatric impairment that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the head and neck
* No other concurrent therapy for the tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-12; Primary Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival
Overall survival
Toxicity
Tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Edward F. McClay, MD, Principal Investigator — San Diego Pacific Oncology & Hematology Associates
Locations (1):
- San Diego Pacific Oncology and Hematology Associates, Incorporated - Encinitas, Encinitas, California, United States